CLINICAL TRIAL: NCT06985394
Title: Vascular Function and Oxidative Stress in Emergency Medical Responders
Acronym: VF-EMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2291409-1
Record Dates: First submitted 2025-02-25; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Function in EMTs
Keywords: EMT; First Responder; Oxidative Stress; Paramedic; Emergency Medical Technician

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antioxidant Supplementation (Experimental): Participants will take two doses of antioxidant supplements in capsule form during their overnight shift: the first dose at 7:00 PM, and the second dose 1.5 hour before their morning vascular function visit (post-shift). Each dose will consist of the following concentrations of antioxidants:
  600 mg of α-lipoic acid, 1,000 mg of vitamin C, and 600 IU of vitamin E.
  Interventions: Dietary Supplement: Antioxidant cocktail
- Placebo Supplementation (Placebo Comparator): Participants will take two doses of placebo supplements in capsule form during their overnight shift: the first dose at 7:00 PM, and the second dose 1.5 hour before their morning vascular function visit (post-shift). Each dose will consist of placebo pills made from microcrystalline cellulose, designed to match the antioxidants in taste, color, and appearance
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Antioxidant cocktail — Participants will take two doses of antioxidant supplements in capsule form during their overnight shift: the first dose at 7:00 PM, and the second dose 1.5 hour before their morning vascular function visit (post-shift). Each dose will consist of the following concentrations of antioxidants:
  600 mg of α-lipoic acid, 1,000 mg of vitamin C, and 600 IU of vitamin E.
  Arms: Antioxidant Supplementation
Dietary Supplement: Placebo — Participants will take two doses of antioxidant supplements in capsule form during their overnight shift: the first dose at 7:00 PM, and the second dose 1.5 hour before their morning vascular function visit (post-shift). Each dose will consist of placebo pills made from microcrystalline cellulose, designed to match the antioxidants in taste, color, and appearance.
  Arms: Placebo Supplementation

SUMMARY:
The goal of this clinical trial is to characterize blood vessel function and oxidative stress (a harmful condition that damages cells and tissues) in emergency medical technicians (EMTs). The main questions it aims to answer are:

1. Does an overnight shift work in emergency medical technicians reduce blood vessel function and increase oxidative stress?
2. Can supplementing with antioxidants help reduce the negative effects of night shift work in emergency medical technicians?

Researchers will compare antioxidants to a placebo (a look-alike substance that contains no drug) to see if antioxidants work in reducing the negative effects of night shift work in emergency medical technicians.

Participants will:

1. Report to the lab two separate times following an overnight shift to assess blood vessel functioning and oxidative stress 3. Take an antioxidant supplement or placebo during each night of shift work.

DETAILED DESCRIPTION:
Heart disease, also referred to as cardiovascular disease, is the leading cause of death worldwide, responsible for about 30% of all deaths. While eating right, staying active, and avoiding cigarettes are key to preventing heart problems, the type of work a person does matters too. Some jobs can negatively affect heart health, especially those with night or irregular shifts. Emergency medical technicians (EMTs), the first responders who help keep our communities safe, often work these challenging schedules.

Shift work means working outside normal business hours-like evenings, nights, and weekends. These irregular schedules, especially overnight shifts, can disrupt the body's natural sleep cycle. This disruption can cause health problems because it goes against the body's internal clock, or circadian rhythm. This rhythm controls important functions like sleep, hormone levels, and heart health. When someone works at night, this clock is disrupted, which can lead to higher stress levels, worse blood vessel function, and even long-term damage to the heart. Research shows that people who work night shifts have a higher risk of heart disease compared to those who work during the day. The risk increases even more the longer someone works night shifts. In fact, studies show that each additional five years of night shift work raises the risk of heart problems by 7%. One night of shift work is all it takes to cause damage to blood vessels and spike stress levels in the body.

This study will examine how night shift work affects emergency medical technicians' heart and blood vessel health. The investigators will compare the function of their blood vessels and levels of oxidative stress (a harmful condition that damages cells and tissues) after working two overnight shifts. To understand how to best help reduce the negative effects of night shift work, this study will also test whether taking antioxidants-substances that protect the body from damage induced by oxidative stress-during one of the shifts can improve blood vessel health and reduce oxidative stress. Emergency medical technicians are a group that have not been researched much in this area and by doing so, this study hopes to learn more about how night shift work affects heart and blood vessel health. If antioxidants can help, this could lead to new ways of protecting shift workers from long-term heart problems-especially emergency medical technicians and first responders, who are vital to our community's safety.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.5 and <35 kg/m²
* Seated resting systolic blood pressure < 140 mmHg, and seated resting diastolic blood pressure < 90 mmHg
* Participant must be an active first responder that works shift work schedules. e.g., emergency medical responders, basic life support emergency medical technicians (i.e., BLS EMT), advanced life support emergency medical technicians (A-EMT), and paramedics
* Participant must have been working shift work for at least 1 year
* Participant must work at least 4 night shifts per month

Exclusion Criteria:

* Participant is unwilling or unable to give consent
* Participant has been diagnosed with any chronic disease (a history of high blood pressure, heart disease, diabetes, cancer, kidney disease)
* Participant has been diagnosed with a sleep disorder (e.g., insomnia, restless leg syndrome, sleep apnea)
* Participant is currently taking melatonin or other sleep aids (e.g., Ambien, sedatives, etc.), or any supplements/medications known to alter sleep patterns. Participants using melatonin must undergo a minimum 72-hour washout period prior to study participation to ensure baseline sleep patterns are not affected[15, 16]
* Resting blood pressure >140/90 mmHg
* Body mass index <18.5 or >35 kg/m2
* Currently pregnant or breast feeding (women only)
* Currently use tobacco or nicotine products (≥1 cigarette, cigar, e-cigarette, vape, or any other nicotine-containing product in the last month), including smokeless tobacco (e.g., chewing tobacco, snuff, dip, snus), nicotine lozenges or gum, heated tobacco products, and any illicit drugs

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Flow Mediated Dilation (FMD) | Visit 2 (1 day)
  Flow-mediated dilation (FMD) is a frequently practiced non-invasive technique which images artery structure and blood flow before, during, and after a period of blood flow occlusion and subsequent increases in blood flow. This creates stress on the inner lining (i.e., endothelium) of the vasculature, inducing a cascade of events which results in relaxation of the smooth muscle surrounding the vessel. Reduced functioning of this mechanism is significantly associated with cardiovascular complications and disease. FMD will be used to assess the diameter and blood flow velocity of the artery located in the upper arm via ultrasonography.
Oxidative Stress | Visit 3 (1 day)
  Electron Paramagnetic Resonance (EPR) Spectroscopy measurements will be conducted using a specialized spectrometer (Bruker EMX Nano) which is designed to detect unpaired electrons in biological samples, a key indicator of oxidative damage. For the EPR procedure, frozen samples of blood plasma will be carefully collected from the participant following standard clinical protocols during their vascular function visits. Briefly, the spin trapping technique will be used where a stabilizing molecule (e.g., spin probe such as cyclic hydroxylamine [CMH]) reacts with the free radical (e.g., superoxide) to form a more stable radical species for analysis (nitroxide). The stable sample will then be placed in the EPR resonator, and the spectrometer will be calibrated using known standards to ensure accurate detection of nitroxide.
Passive Leg Movement (PLM) | Visit 2 (1 day)
  PLM is a newer, non-invasive method of assessing vascular function that is also mediated through the responsiveness of the endothelium. This assessment may provide additional insight on vascular function specific to the lower extremity. Briefly, participants will have one minute of blood flow velocity of the right femoral artery recorded (distal to inguinal crease, proximal to deep and superficial bifurcation) via Doppler ultrasound, while sitting with back upright, both legs supported, and knees fully extended (i.e., 180 degrees). Passive movement will then be initiated by a second team member who will continuously move the participant's right leg through 90 degrees of motion for two minutes. Participants will be urged to remain passive and to avoid any assistance with limb motion. Blood flow velocity of the right femoral artery will be continuously recorded during the entire 3 minute test to investigate changes in blood flow velocity during passive leg movement.
Flow Mediated Dilation (FMD) | Visit 3 (1 day)
  Flow-mediated dilation (FMD) is a frequently practiced non-invasive technique which images artery structure and blood flow before, during, and after a period of blood flow occlusion and subsequent increases in blood flow. This creates stress on the inner lining (i.e., endothelium) of the vasculature, inducing a cascade of events which results in relaxation of the smooth muscle surrounding the vessel. Reduced functioning of this mechanism is significantly associated with cardiovascular complications and disease. FMD will be used to assess the diameter and blood flow velocity of the artery located in the upper arm via ultrasonography.
Passive Leg Movement (PLM) | Visit 3 (1 day)
  PLM is a newer, non-invasive method of assessing vascular function that is also mediated through the responsiveness of the endothelium. This assessment may provide additional insight on vascular function specific to the lower extremity. Briefly, participants will have one minute of blood flow velocity of the right femoral artery recorded (distal to inguinal crease, proximal to deep and superficial bifurcation) via Doppler ultrasound, while sitting with back upright, both legs supported, and knees fully extended (i.e., 180 degrees). Passive movement will then be initiated by a second team member who will continuously move the participant's right leg through 90 degrees of motion for two minutes. Participants will be urged to remain passive and to avoid any assistance with limb motion. Blood flow velocity of the right femoral artery will be continuously recorded during the entire 3 minute test to investigate changes in blood flow velocity during passive leg movement.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared as this study is only being conducted at one location.